CLINICAL TRIAL: NCT06522750
Title: Pilot Study on the Feasibility of an RCT: Evaluating Periodic Fasting as a Treatment Strategy for Long Covid in Adults
Brief Title: Periodic Fasting for Treatment of Long Covid in Adults: a Pilot Study
Acronym: FASTCOV-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202401/03
Record Dates: First submitted 2024-05-17; First posted 2024-07-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Long Covid; Chronic Inflammation
Keywords: long covid; fasting; caloric restriction; chronic inflammation; dysbiosis; mitochondrial dysfunction; thrombosis
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fasting; Dysbiosis; Mitochondrial Diseases; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 participants. Long covid patients. (Experimental): All patients will undergo a caloric restriction diet for a week.This begins with the intake of a laxative fluid on the first fasting day. This fluid aids in bowel emptying, akin to preparations for a colonoscopy. Detailed instructions on how to use it will be provided along with the laxative, and the study physician or dietary team will discuss dosage and intake with you. The caloric restriction period will last for 7 days and then be broken with the consumption of an apple. Following the breaking of the fast, three build-up days will follow to gradually increase food intake.
  Interventions: Other: 7-day ambulatory caloric restriction intervention using the Buchinger-Wilhelmi method

INTERVENTIONS:
Other: 7-day ambulatory caloric restriction intervention using the Buchinger-Wilhelmi method — Buchinger-Wilhelmi method, will be administered in an ambulatory setting under physician guidance. It involves an initial bowel cleanse followed by 7-day fasting period. The initial bowel cleanse will be performed according to the standard procedure commonly used for colonoscopy preparation. During the fasting period, subjects will be provided with a dietary energy supply of a maximum of 350 kcal per day, primarily consisting of vegetable broths as well as fresh vegetable juices. Patients will only be allowed to consume calorie-free and unsweetened water or tea in addition to the prescribed diet.

SUMMARY:
Background:

Long COVID, characterized by persistent symptoms following acute COVID-19 infection, has emerged as a significant public health concern. Symptoms range from fatigue, cognitive impairments, to respiratory difficulties, affecting patients' quality of life. Dietary interventions, particularly fasting, have historically been used to modulate immune responses and improve health outcomes in various conditions. The Buchinger-Wilhelmi method represents a structured and medically supervised fasting approach. Given the inflammatory nature of long COVID, fasting may offer therapeutic benefits by modulating the immune response, enhancing cellular repair mechanisms, and resetting metabolic processes.

Objectives:

This clinical trial aims to assess the feasibility of a 7-day ambulatory fasting intervention using the Buchinger-Wilhelmi method on long COVID patients as primary objective. As secondary objectives, the study will investigate the potential beneficial impact of fasting on clinical, biological, and psychological parameters over a period of 4 weeks, offering insights into potential therapeutic avenues for long COVID management.

Study timeline:

The research will span a period of 4 weeks

Study population:

This study aims to recruit around 20 participants, who will all receive a fasting intervention using the Buchinger-Wilhelmi method.

Biological sample and data collection:

Participants will undergo various data and sample collection procedures, including blood draws of up to 90 42 ml per visit, collection of peripheral mononuclear cells, stool samples, and completion of questionnaires in a smartphone-based Application (MyCap).

Sample analysis:

The collected samples will be subjected to a range of analyses, including the assessment of serological markers for routine blood chemistry, evaluation of inflammation markers, and examination of stool samples.

DETAILED DESCRIPTION:
Background Long COVID syndrome (LCS) is a heterogeneous clinical condition that develops after acute SARS-CoV-2 infection, affecting at least 10% of patients. LCS is characterized by persistent symptoms lasting longer than 2-3 months following a confirmed SARS-CoV-2 infection. The most disruptive symptoms include fatigue, shortness of breath, pain, depression/anxiety, and cognitive impairment, significantly impacting daily activities, income, and quality of life.

Pathophysiology of LCS

Immunological Dysregulation:

Persistent activation of monocyte populations, including resident and infiltrating macrophages, dendritic cells, and neutrophils, potentially causing tissue damage.

Reservoirs of SARS-CoV-2 may persist, particularly in respiratory and gastrointestinal tracts, contributing to ongoing lymphocyte activation.

Autoimmunity involving T-cells and B-cells has been observed, with cytokines such as interferon gamma, IL-2, IL-4, IL-6, IL-8, IL-10, and IL-17 frequently implicated.

Tissue fibrosis, a consequence of inflammation, is commonly reported.

Vascular Dysfunction and Coagulopathy:

Impaired fibrinolysis and platelet hyperactivation contribute to microclot formation, entrapping pro-inflammatory molecules like IL-6.

Platelet-poor plasma in LCS patients shows high levels of fibrin amyloid microclots, impairing microcirculation and exacerbating immunopathology.

Aberrant immune cell activity increases thrombosis through autoantibodies and NETosis.

Persistent endothelial dysfunction is a common feature, contributing to numerous LCS symptoms.

Gastrointestinal Involvement:

SARS-CoV-2 infection reduces intestinal microbiota diversity, with recovery correlating to reduced LCS risk.

Specific bacterial taxa, such as Escherichia, are associated with severe COVID-19 and LCS.

Functional dyspepsia and irritable bowel syndrome, related to microbial dysbiosis, are common post-COVID conditions.

Gut microbiota influences LCS-related biological functions, particularly psychological symptoms, through modulation of brain chemicals and gut-blood barrier disruption.

Potential of Fasting as a Treatment for LCS Fasting shows promise as a treatment for LCS by modulating the same cellular systems affected by LCS. A recent small study indicated that 92% of LCS patients experienced symptom improvement during long-term fasting, with notable effects on circulating inflammatory molecules, C-reactive protein levels, and dyslipidemia. Fasting can increase beneficial gut microbial genera and alter blood metabolites, potentially disrupting dysfunctional circuits in LCS.

Significance LCS affects over 150 million people worldwide, with more than half experiencing significant work and lifestyle disruptions. Effective, low-cost, and attainable therapeutic options are urgently needed. Medically supervised fasting, particularly intermittent fasting, could be an accessible and safe intervention with minimal physician oversight and low malnutrition risk. Fasting may also prevent other chronic illnesses associated with LCS, such as type 2 diabetes mellitus.

Hypothesis Our primary hypothesis is that ambulatory fasting intervention using the Buchinger-Wilhelmi method is a feasible treatment for LCS. We propose that medically supervised long-term fasting will improve perceived health and quality of life in LCS patients by disrupting inflammatory immuno-metabolic feed-forward loops, thus ameliorating immune and vascular pathologies.

Methodology and Analysis Patient Eligibility

Inclusion Criteria:

Age 18-64 Diagnosis of LCS (post-acute COVID-19 symptoms persisting ≥12 weeks) Normal BMI (18.5 to 25 kg/m²) Marginal iron status (PF < 25 ng/ml) Ability to communicate in and comprehend English, German, or French Written and signed consent Willingness to consent to specimen collection and use

Exclusion Criteria:

BMI < 18.5 kg/m² or significant recent weight loss History of eating disorders within the past five years Severe internal disease or chronic inflammatory illness other than LCS Participation in another intervention study Recent fasting or vegan diet Pregnancy or breastfeeding Existing ME/CFS or early autonomous dysfunction Chronic inflammatory bowel diseases, celiac disease, or colorectal cancer Use of anti-psychotic drugs or recent antibiotic use Contraindication for additional blood draws Start of novel drug therapy Intervention

The primary goal is to perform a single period of periodic fasting (PF) using the Buchinger procedure, involving an initial bowel cleanse followed by a 7-day fasting period. The fasting regimen includes:

Preparation Phase: Three days of relief with reduced food intake, avoiding stimulants.

Fasting Week: A laxative fluid intake on the first day, followed by 7 days of a dietary energy supply of a maximum of 350 kcal per day (vegetable broths and juices), and consumption of calorie-free water or tea.

Support and Guidance: Detailed instructions, face-to-face consultations, and digital application (MyCap) for adherence confirmation via urine ketone measurements.

Sample and Data Collection Sample Size: 20 patients for the pilot study to test feasibility.

Study Outline:

Inclusion visit for risk explanation, medical history, and physical examination.

Daily follow-up via telephone and online appointments during the fasting phase. Questionnaire-based assessment via MyCap Smartphone Application.

Parameters to be Quantified:

Blood samples for safety parameters, metabolites, immune activity indicators, and additional analyses.

Stool samples for microbiome composition and activity. Urine samples for metabolomics. Saliva samples for cortisol measurements. Analysis and Results Interpretation Results will be analyzed descriptively, with means, standard deviations, and graphs summarizing data. Exploratory analysis will identify patterns, trends, or unexpected results. Correlation with improvement in biomedical parameters will be assessed, with a larger study needed for establishing causal links.

Risks Blood Draw: Discomfort, bleeding, swelling, pain, rare nerve damage, or infection at the injection site, and fainting risk.

Periodic Fasting Protocol: Reduction in blood pressure, closely monitored with non-medical interventions if necessary.

Data Collection and Storage Data is collected using REDCap, a secure, web-based software platform, with pseudonymized data stored for at least 10 years post-study. The Principal Investigator ensures compliance with national laws and GDPR.

Regulatory and Ethical Considerations Informed Consent: Participants receive an easily understood Participant Information Sheet and Informed Consent Form, with contact information for study personnel.

Confidentiality and Privacy: Compliance with national laws and GDPR, with pseudonymized data transfer to third parties only with participant consent.

Financing and Insurance: Supported by the Direction de la Santé, CHNP, and the University of Luxembourg.

Conclusion This pilot study aims to test the feasibility of using the Buchinger-Wilhelmi fasting method for treating LCS. If successful, fasting could provide a low-cost, accessible, and effective therapeutic option for LCS sufferers worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Diagnosis Long Covid Syndrome (post-acute COVID-19 symptoms persisting ≥12 weeks)
* Normal body Mass Index (18.5 to 25 kg/m2)
* Marginal Iron status ( PF< 25 ng/ml)
* Able to communicate in and comprehend English and/or German and/or French language
* Present written / signed declaration of consent
* Ability to understand the patient information and willingness to sign the consent form
* Consent to specimen collection and specimen use

Exclusion Criteria:

* Current underweight condition (body mass index less than 18.5 kg/m2) or weight loss exceeding 3 kg within the last month or 5 kg within the last three months.
* Existing / current eating disorder within the past five years (e.g., anorexia, bulimia).
* Psychiatric condition that limits understanding of the examination protocol (unable to consent)
* Severe internal disease (e.g. kidney deficiency with creatinine > 2mg/dl), chronic inflammatory illness other than LCS
* Participation in another intervention study.
* Existing vegan diet or fasting during the last six months
* Pregnancy or breastfeeding status.
* Presence or suspicion of pre-existing ME/CFS or early autonomous dysfunction
* Diagnosis of chronic inflammatory bowel diseases, celiac disease or colorectal cancer according to the guidelines of the German Society of Gastroenterology
* Use of anti-psychotic drugs
* Antibiotic use during the previous 12 months
* Start of novel drug therapy
* Contraindication for additional blood draws (e.g. hemoglobin <10)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional protocol | 4 weeks
  Patient's level of health and wellbeing from a nutritional point of view
Fatigue assessment Scale (FAS) | 4 weeks
  Level of fatigue through three factors (General Fatigue, Physical Fatigue and Concentration/Motivation).
Quality of Life (WHOQOL) | 4 weeks
  Quality of Life as an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns.
Functionality (WHODAS 2.0) | 4 weeks
  Impact of Long Covid in terms of functioning.
Anxiety (GAD-7) | 4 weeks
  Generalized anxiety disorder in the last 2 weeks
Depression (PHQ-9) | 4 weeks
  Presence and severity of depressive symptoms
Mood States | 4 weeks
  Transient fluctuating moods or affective states
Blood preasure | 4 weeks
  Force or pressure of blood on the arteries when the heart is pumping

SECONDARY OUTCOMES:
Urine Metabolomics | 4 weeks
  Metabolites in urine
Gut Microbiome | 4 weeks
  Microbiota in stool
Stool Metabolomics | 4 weeks
  Metabolites in stool
Blood cytokines | 4 weeks
  Cytokines using Quanterix technology
Blood Mitochondrial dysfunction | 4 weeks
  Mitochondrial cell-free DNA
Blood Epigenetics | 4 weeks
  Methylation profiling microarray
Blood test | 4 weeks
  Metabolites in blood

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Gomez Bravo, PhD, Principal Investigator — Rehaklinik du Centre Hospitalier Neuro-Psychiatrique (CHNP), UL
Locations (1):
- Rehaklinik CHNP, Ettelbruck, Luxembourg